## **DEPARTMENT OF PSYCHIATRY**

NEUROSCIENCES BUILDING WARNEFORD HOSPITAL OXFORD OX3 7JX, U.K. www.psych.ox.ac.uk





1

<u>Principal Investigator</u>: Dr Susannah Murphy <u>Email</u>: susannah.murphy@psych.ox.ac.uk

**Tel**: +44 (0)1865 618313

**Primary Researcher**: Michael Colwell, DPhil Student

Tel: +44 (0)1865 618 303

Email: michael.colwell@psych.ox.ac.uk

## Consent to take part in 'An fMRI investigation of the effects of selective histamine-3 antagonism on cognitive and emotional processing in healthy individuals'

CUREC Approval Reference: R83940/RE001

Purpose of Study: To investigate the effects of pitolisant on emotional processing and cognitive ability, comparing the effects of the drug with placebo.

| | | Please initial each |
|---|---|---|
| 1 | I confirm that I have read and understand the information sheet version dated for the above research. I have had the opportunity to consider the information carefully, ask questions and have had these questions answered satisfactorily. | |
| 2 | I understand that my participation is voluntary and that I am free to withdraw at any point until <b>01/12/2023</b> , without giving any reason. | |
| 3 | I have been advised about the potential risks associated with taking part in this research and have taken these into consideration before consenting to participate. | |
| 4 | I have been advised as to what I need to do for this research (especially with regard to pitolisant intake) and I agree to follow the instructions given to me. | |
| 5 | To the best of my knowledge, I do not meet any of the exclusion criteria outlined in the information sheet for this research. If this changes at a later date during study participation, I agree to notify the researchers immediately. | |
| 6 | I understand that data collected and scans during the study may be looked at by designated individuals from the University of Oxford. I give permission for these individuals to access my data. | |
| 7 | I understand who will have access to personal data provided, how the data will be stored and what will happen to the data at the end of the project. | |
| 8 | I understand that I will not be identifiable from any research publications, presentations or doctoral theses. | |
| 9 | I understand that the MRI scans in this study are for research and they are not useful for medical diagnosis, and that scans are not routinely looked at by a doctor. If a concern is raised about a possible abnormality on my scan, I will be informed if a doctor thinks this is medically important such that the finding has | |

clear implications for my current or future health.

| 10 | I understand how this research will be written up and published. | | |
|---|---|---|---|
| 11 | I understand that research data collected in this study may be shared with other researchers, including those working outside of the UK and the EU, via means including an online repository. I understand that it will be shared in a form that does not identify me. | | |
| 12 | I understand that this project has been reviewed by, and received ethics clearance through, the University of Oxford Central University Research Ethics Committee. | | |
| 13 | I understand how to raise a concern or make a complaint. | | |
| 14 | I agree to take part in the study. | | |
| Name of | Participant | dd / mm / yyyy<br>Date | Signature |
| Name of | person taking consent | dd / mm / yyyy<br>Date | <br>Signature |